CLINICAL TRIAL: NCT02270333
Title: Effects of Inspiratory Muscle Training in Patients With Sarcoidosis
Brief Title: Inspiratory Muscle Training in Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GaziU
Record Dates: First submitted 2014-10-08; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; inspiratory muscle strength; exercise capacity; quality of life
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Intervention: Treatment group received inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device .
  Interventions: Device: Inspiratory muscle training
- Control group (Sham Comparator): Sham: Control group received sham inspiratory muscle training using POWERbreathe Classic threshold loading device .
  Interventions: Device: Sham inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Treatment group received inspiratory muscle training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 40% of maximal inspiratory pressure (MIP).
  The MIP was measured at supervised session each week, and 40% of measured MIP value was the new training workload.
  The treatment group trained for 30 min-per/day, 7 days/week, for 6 weeks. Six sessions at home and 1 session were performed at department.
  Arms: Treatment group
Device: Sham inspiratory muscle training — Control group received sham inspiratory muscle training (IMT) at fixed workload, 5% of MIP using threshold loading device (POWERbreathe Classic device IMT Technologies Ltd. Birmingham, England).
  The control group trained for 30 min-per/day, 7 days/week, for 6 weeks. Six sessions at home and 1 session were performed at department.
  Arms: Control group

SUMMARY:
Respiratory muscle weakness results with decreased exercise capacity, worse fatigue, dyspnea and quality of life in patients with sarcoidosis. However, no study investigated the effects of inspiratory muscle training (IMT), therefore effects of IMT on outcomes in patients with sarcoidosis were investigated.

DETAILED DESCRIPTION:
Patients were diagnosed with sarcoidosis according to the criteria of the latest American Thoracic Society (ATS)/European Respiratory Society (ERS)/World Association of Sarcoidosis and Other Granulomatous (WASOG) Disorders statement on sarcoidosis. Primary outcome measurement was respiratory muscle strength, secondary outcomes were, exercise capacity quality of life, fatigue and depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Under standard medication
* Stage I and IV
* No change in medications over three months

Exclusion Criteria:

* Cognitive disorders
* Current corticosteroid use
* Having co-morbidity to prevent performing IMT
* Acute infection
* Orthopedic and neurological problems

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory and expiratory muscle strength (MIP, MEP) | 6 weeks
  Mouth pressure device

SECONDARY OUTCOMES:
Exercise Capacity | 6 weeks
  Six-minute walk test (6MWT)
Maximal Exercise Capacity | 6 weeks
  Modified incremental shuttle walk test (ISWT)
Fatigue | 6 weeks
  Fatigue Severity Scale (FSS)
Pulmonary function and diffusing capacity | 6 weeks
  Spirometry
Peripheral muscle strength | 6 weeks
  Hand-held dynamometer
Dyspnea | 6 weeks
  Modified Borg and Modified Medical Research Council (MMRC) dyspnea scales
Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS))
Quality of life | 6 weeks
  Saint George's Respiratory Questionnaire (SGRQ) (Turkish versions of all scales)

CONTACTS AND LOCATIONS:
Overall Officials: Müşerrefe Nur Karadallı, MSc., Study Chair — Gazi University; Burcu Camcıoğlu, MSc., Principal Investigator — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Nurdan Köktürk, MD, Principal Investigator — Gazi University; Haluk Türktaş, MD, Principal Investigator — Gazi University

REFERENCES:
- [Result] Spruit MA, Thomeer MJ, Gosselink R, Troosters T, Kasran A, Debrock AJ, Demedts MG, Decramer M. Skeletal muscle weakness in patients with sarcoidosis and its relationship with exercise intolerance and reduced health status. Thorax. 2005 Jan;60(1):32-8. doi: 10.1136/thx.2004.022244. PMID 15618580
- [Result] Kabitz HJ, Lang F, Walterspacher S, Sorichter S, Muller-Quernheim J, Windisch W. Impact of impaired inspiratory muscle strength on dyspnea and walking capacity in sarcoidosis. Chest. 2006 Nov;130(5):1496-502. doi: 10.1378/chest.130.5.1496. PMID 17099029
- [Result] Baydur A, Alsalek M, Louie SG, Sharma OP. Respiratory muscle strength, lung function, and dyspnea in patients with sarcoidosis. Chest. 2001 Jul;120(1):102-8. doi: 10.1378/chest.120.1.102. PMID 11451823
- [Result] Wirnsberger RM, Drent M, Hekelaar N, Breteler MH, Drent S, Wouters EF, Dekhuijzen PN. Relationship between respiratory muscle function and quality of life in sarcoidosis. Eur Respir J. 1997 Jul;10(7):1450-5. doi: 10.1183/09031936.97.10071450. PMID 9230229
- [Derived] Karadalli MN, Bosnak-Guclu M, Camcioglu B, Kokturk N, Turktas H. Effects of Inspiratory Muscle Training in Subjects With Sarcoidosis: A Randomized Controlled Clinical Trial. Respir Care. 2016 Apr;61(4):483-94. doi: 10.4187/respcare.04312. Epub 2015 Dec 29. PMID 26715771